CLINICAL TRIAL: NCT02841033
Title: A Phase I-II Trial of Daratumumab for the Treatment of Patients With AL Amyloidosis
Brief Title: Daratumumab for the Treatment of Patients With AL Amyloidosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-35360; 54767414AMY2002 (Other: Janssen Pharmaceuticals)
Record Dates: First submitted 2016-06-14; First posted 2016-07-21 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: AL Amyloidosis
Keywords: Daratumumab
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daratumumab (Experimental): Daratumumab, 16mg/kg body weight in 1000 mL for the first dose, followed by 500mL for subsequent doses, once weekly for two months, then every 2 weeks for four months, then once each month.
  Interventions: Drug: daratumumab

INTERVENTIONS:
Drug: daratumumab — Daratumumab by IV infusion once weekly for two months, then every 2 weeks for four months, then once each month until progression or inability to tolerate.
  Other Names: Darzalex

SUMMARY:
Participants with AL Amyloidosis will receive the drug daratumumab by IV infusion once weekly for two months, then every 2 weeks for four months, then once each month. Study treatment may continue until disease progression, unacceptable toxicity, or decision to withdraw from the trial. Disease evaluations will be performed every three months until disease progression.

DETAILED DESCRIPTION:
This Phase I/II study is intended to evaluate the safety and tolerability of infusion of daratumumab in AL amyloidosis, specifically with respect to infusion reactions. In addition, the investigators would like to assess organ response with respect to cardiac biomarkers and proteinuria, as well as hematologic response and time to next treatment. Participants with AL Amyloidosis will receive the drug daratumumab by IV infusion once weekly for two months, then every 2 weeks for four months, then once each month. Study treatment may continue until disease progression, unacceptable toxicity, or decision to withdraw from the trial. Disease evaluations will be performed every three months until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of primary systemic (AL) amyloidosis:

  1. At least one tissue demonstrating positive Congo Red staining with characteristic apple green birefringence AND
  2. Evidence of a clonal plasma cell dyscrasia:

  i. Monoclonal protein in the serum and/or urine by immunofixation electrophoresis AND/OR ii. Abnormal serum free light chain assay AND/OR iii. Clonal plasma cell population in the bone marrow demonstrated by immunohistochemistry, flow cytometry or in situ hybridization AND

  c. Evidence of organ involvement other than carpal tunnel syndrome. Confirmation of tissue diagnosis at all sites of organ dysfunction is encouraged, but not required.
* Must have relapsed after or been refractory to at least one prior treatment regimen of proven efficacy in the treatment of AL amyloidosis
* Must be > 18 years of age.
* Must have a performance status of 0-2 by Eastern Cooperative Oncology Group (ECOG) criteria
* Must have adequate hepatic function as evidenced by serum bilirubin values < 2.0 mg/dL; alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) < 3x upper limit of normal (ULN).
* Must have an absolute neutrophil count ≥1000/mm3, hemoglobin ≥7.5 g/dL, and platelet count ≥50×109/L

Exclusion Criteria:

* • Renal Insufficiency (CrCL <20mL/min), calculated by Cockcroft-Gault Equation Creatinine Clearance = Sex * ((140 - Age) / (SerumCreat)) * (Weight / 72) Equation parameters such as sex have two or more discrete values that may be used in the calculation. The numbers in the parentheses, e.g. (1), represent the values that will be used. The default unit of measure for weight is kilograms. Please verify that the correct unit of measure has been selected.

  * Mayo clinic cardiac biomarker stage IIIb
  * Evidence of significant cardiovascular conditions as specified below:
* B-type Natriuretic Peptide; N-terminal pro b-type Natriuretic Peptide (NT-ProBNP) > 8500 ng/L (Mayo Stage IIIb patients are excluded)
* New York Heart Association (NYHA) classification IIIB or IV heart failure
* Unstable Angina, Arrhythmia, prolonged corrected QT (QTc) interval, symptomatic orthostatic hypotension, or supine systolic blood pressure < 90 mm Hg.
* left ventricular ejection fraction (LVEF) <40%

  * Overt multiple myeloma (>30% bone marrow plasmacytosis, extensive (>2) lytic lesions, or hypercalcemia).
  * Plan for autologous stem cell transplant in the six months prior to study drug (stem cell collection is permitted during the first six months of study treatment)
  * Any form of secondary or familial (ATTR) amyloidosis
  * The presence or history of another malignancy is not allowed except for the following:

    * adequately treated basal cell or squamous cell skin cancer,
    * in situ cervical cancer,
    * adequately treated Stage I or II cancer from which the patient is currently in complete remission, any other cancer from which the patient has been disease-free for 5 years.
  * Known to be Human Immunodeficiency Virus (HIV) positivity.
  * Pregnant or nursing women. Women and men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
  * Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume at one second (FEV1) <50% of predicted normal. Note that forced expiratory volume at one second FEV1 testing is required for patients suspected of having COPD.
  * Known moderate or severe persistent asthma within the past 2 years or currently has uncontrolled asthma of any classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaishali Sanchorawala, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchorawala V, Sarosiek S, Schulman A, Mistark M, Migre ME, Cruz R, Sloan JM, Brauneis D, Shelton AC. Safety, tolerability, and response rates of daratumumab in relapsed AL amyloidosis: results of a phase 2 study. Blood. 2020 Apr 30;135(18):1541-1547. doi: 10.1182/blood.2019004436. PMID 31978210
- See also: creatinine clearance cockcroft-gault formula — http://reference.medscape.com/calculator/creatinine-clearance-cockcroft-gault

RESULTS

PARTICIPANT FLOW:
Groups:
- Daratumumab: Daratumumab, 16mg/kg body weight in 1000 mL for the first dose, followed by 500mL for subsequent doses, once weekly for two months, then every 2 weeks for four months, then once each month for up to 24 total cycles.
  Daratumumab: Daratumumab by IV infusion once weekly for two months, then every 2 weeks for four months, then once each month until progression, inability to tolerate, or 24 cycles completed.
Period: Overall Study
Arm/Group | Daratumumab
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Daratumumab
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 63 [42 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 16
  Black or African American | 7
  Asian | 0
  Hispanic or Latino | 2
  Other | 0
Region of Enrollment [Number; unit: participants]
  United States | 22
Time since initial diagnosis [Median (Full Range); unit: months] | 48 [8 to 184]
Prior therapies [Median (Full Range); unit: lines of treatment] | 2 [1 to 7]
Time since last plasma cell-directed treatment [Median (Full Range); unit: months] | 9 [1 to 180]
dFLC [Median (Full Range); unit: mg/L] | 80.7 [2.9 to 854]
Number of organ systems involved [Median (Full Range); unit: organ systems] | 2 [1 to 5]
NYHA Class II or III [Count of Participants; unit: Participants] — The NYHA [New York Heart Association} classification of heart failure uses categories I, II, III, and IV for patients' symptoms. The higher the Class, the more symptoms of heart failure that the patient has. Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.
  Participants | 11

OUTCOME MEASURES:

1. Primary Outcome: Assess the Number of Patients Who Respond to Treatment
Description: Number of participants with response and ability to tolerate study treatment in each of these categories: Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD).
  All participants were able to tolerate study treatment.
  Per protocol, overall response designations are a combination of hematologic response.
  A CR is defined as negative serum and urine immunofixation electrophoresis with normal serum free light chain ratio; a VGPR is reduction in the dFLC* to <40 mg/L, a PR is dFLC reduction by >50%; SD is not meeting criteria for CR, VGPR, PR, or PD; and PD is an increase in FLC of 50% to >100 mg/L.
  * "dFLC" is difference in involved and uninvolved serum Free Light-Chain levels.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 22
Participants
  Complete Response (CR) | 5
  Very Good Partial Response (VGPR) | 13
  Partial Response (PR) | 2
  Stable Disease (SD) | 1
  Progressive Disease (PD) | 1

2. Secondary Outcome: Time to Next Treatment
Description: Number of months from study drug initiation to starting another treatment
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 22
Participants
  <12 months | 3
  >12 months | 1
  No further treatment | 18

3. Secondary Outcome: Assess Hematologic Response Based on Blood and Urine Testing Using Standard Criteria
Description: Number of patients with hematologic complete response (CR), very good partial response (VGPR), or partial response (PR).
  Per protocol, a hematologic CR is defined as negative serum and urine immunofixation electrophoresis with normal serum free light chain ratio; a VGPR is reduction in the dFLC* to <40 mg/L; and a PR is dFLC reduction by >50%.
  * "dFLC" is difference in involved and uninvolved serum free light-chain levels
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 22
Participants
  Complete Response, Very Good Partial Response, or Partial Response | 20
  Stable Disease or Progressive Disease | 2

4. Secondary Outcome: Assess Organ Responses Based on Standard Criteria Included in Protocol
Description: Number of patients with organ response based on standard criteria included in protocol.
  Cardiac response is defined as: NT-proBNP response (>30% and >300 ng/L decrease in patients with a baseline NT-proBNP >650 ng/L; and/or NYHA class response (> two-class decrease if baseline NYHA class 3 or 4)
  Renal response is defined as: Decrease in proteinuria by > 30% or below 0.5 g/24 h without renal progression. Serum creatinine and creatinine clearance must not worsen by 25% over baseline
Time Frame: 3 months
Population: 19 evaluable patients with cardiac and/or renal involvement.
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 19
Participants | 14

ADVERSE EVENTS:
Time Frame: First day of treatment through the end of treatment visit. Duration of subject treatment varied from 2 months to 24 months.
Description: Adverse events were assessed at every study treatment visit.
Arm/Group | Daratumumab
All-Cause Mortality (participants affected / at risk) | 4/22
Serious Adverse Events (participants affected / at risk) | 11/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daratumumab (N=22)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 4 (5)
CK increased (Investigations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
CPK increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Gastrointestinal hemorrhage - melena (Gastrointestinal disorders) | 1 (1)
Heart failure (Cardiac disorders) | 3 (5)
Hematuria (Renal and urinary disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Myocardial infarction (NSTEMI) (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Renal and urinary disorders - other, UTI sepsis (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Syncope (Nervous system disorders) | 2 (3)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Urine output decreased (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daratumumab (N=22)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 3 (6)
Palpitations (Cardiac disorders) | 2 (5)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Hearing loss (Ear and labyrinth disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Endocrine disorder - other, specify: TSH elevated (Endocrine disorders) | 3 (10)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 1 (2)
Blurred vision (Eye disorders) | 3 (3)
Cataract (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 2 (2)
Eye disorders - other, specify: cloudiness (Eye disorders) | 1 (2)
Eye disorders - other, specify: obstructive tear duct (Eye disorders) | 1 (1)
Eye disorders - other, specify: redness (Eye disorders) | 1 (1)
Eye disorders - other, specify: scleral abrasian (Eye disorders) | 1 (3)
Eye disorders - other, specify: Scotoma (Eye disorders) | 1 (10)
Eye disorders - other, specify: subconjunctival hemorrhage (Eye disorders) | 7 (10)
Eye infection (Eye disorders) | 1 (1)
Floaters (Eye disorders) | 1 (4)
Watering eyes (Eye disorders) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 7 (16)
Abdominal pain (Gastrointestinal disorders) | 8 (10)
Anal hemorrhage (Gastrointestinal disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (16)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 19 (68)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal Reflux (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorder - other, specify: inguinal hernia (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorder - other, specify: black stool (Gastrointestinal disorders) | 1 (2)
Gastrointestinal disorder - other, specify: broken tooth (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder - other, specify: H. pylori (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder - other, specify: Tooth extraction (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorder - other, specify: ulcer - Left lateral tongue (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder - other, specify: viral gastroenteritis (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 13 (35)
Oral pain (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 8 (11)
Chest pain (General disorders) | 1 (5)
Chest pain - cardiac (General disorders) | 1 (1)
Chest pain - non cardiac (General disorders) | 1 (2)
Chills (General disorders) | 4 (4)
Edema limbs (General disorders) | 10 (12)
Fatigue (General disorders) | 16 (33)
Fever (General disorders) | 7 (10)
Flu like symptoms (General disorders) | 2 (3)
Gait disturbance (General disorders) | 1 (2)
Localized Edema (General disorders) | 3 (4)
Immune system disorders - other, specify: lymphadenopathy (Immune system disorders) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 8 (17)
Sinusitis (Infections and infestations) | 3 (3)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 11 (21)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 10 (14)
Fall (Injury, poisoning and procedural complications) | 2 (6)
Alanine aminotransferase increased (ALTT) (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 10 (24)
Anemia (Investigations) | 15 (42)
Anorexia (Investigations) | 1 (1)
Aspartate aminotransferase increased (AST) (Investigations) | 8 (18)
Cardiac troponin I increased (Investigations) | 10 (30)
Cholesterol high (Investigations) | 13 (32)
CPK increased (Investigations) | 10 (31)
Creatinine Increased (Investigations) | 17 (67)
Cystitis non-infective (Investigations) | 1 (1)
Investigations - other, specify: Lactate dehydrogenase elevated (Investigations) | 2 (3)
Lymphocyte count decreased (Investigations) | 18 (76)
Neutrophil count decreased (Investigations) | 5 (14)
Platelet count decreased (Investigations) | 10 (18)
Serum amylase increased (Investigations) | 2 (2)
Total bilirubin increased (Investigations) | 6 (27)
Weight gain (Investigations) | 2 (2)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 6 (11)
Anorexia (Metabolism and nutrition disorders) | 7 (13)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 14 (23)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 16 (61)
Hyperuricemia (Metabolism and nutrition disorders) | 13 (26)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (27)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (8)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 7 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (29)
Metabolic and nutrition disorders - other, specify: increased appetite (Metabolism and nutrition disorders) | 2 (2)
Metabolic and nutrition disorders - other, specify: iron deficiency (Metabolism and nutrition disorders) | 8 (9)
Metabolic and nutrition disorders - other, specify: Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Metabolic and nutrition disorders - other, specify: vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (3)
Arthalgia (Musculoskeletal and connective tissue disorders) | 7 (12)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (28)
Fever (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal and connective tissue disorder - other, specify: Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - other, specify: Restless legs (Musculoskeletal and connective tissue disorders) | 4 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (41)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (15)
Neck stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (15)
Neoplasms - other, specify: basal cell carcinoma on sternum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 11 (24)
Dysgeusia (Nervous system disorders) | 2 (2)
Dysphagia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 14 (47)
Memory impairment (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify: Autonomic Postural Hypotension (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 8 (15)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (forgetfullness) (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 12 (15)
Irritability (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 11 (30)
Hematuria (Renal and urinary disorders) | 5 (8)
Nocturia (Renal and urinary disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 5 (6)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (2)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (46)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (15)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 7 (13)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 10 (19)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Nail infection (Skin and subcutaneous tissue disorders) | 2 (2)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (9)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (5)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 7 (18)
Skin & subcutaneous tissue disorders - other, specify: cercarial dermatitis/swimmer's itch (Skin and subcutaneous tissue disorders) | 1 (4)
Skin and Subcutaneous tissue disorders - other, specify: Abrasion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and Subcutaneous tissue disorders - other, specify: bug bite (Skin and subcutaneous tissue disorders) | 3 (4)
Skin and Subcutaneous tissue disorders - other, specify: erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and Subcutaneous tissue disorders - other, specify: Laceration (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders - other, specify: Skin sensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and Subcutaneous tissue disorders - other, specify: Wound (Skin and subcutaneous tissue disorders) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical procedure - other, specify: Biopsy /wart removal (Surgical and medical procedures) | 1 (1)
Surgical procedure - other, specify: biopsy, face, head, back (Surgical and medical procedures) | 1 (1)
Surgical procedure - other, specify: pre-cancerous areas removed (Surgical and medical procedures) | 2 (3)
Surgical procedure - other, specify: shaved excision of dysplastic nevus (Surgical and medical procedures) | 1 (1)
Arterial injury (Vascular disorders) | 1 (2)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT02841033/Prot_SAP_000.pdf